CLINICAL TRIAL: NCT02660502
Title: A Double-blind, Comparator-controlled, Randomised, Three-period Crossover Euglycemic Clamp Trial to Evaluate Pharmacokinetics of Single Doses of BioChaperone Insulin Lispro in Healthy Japanese Subjects
Brief Title: An Euglycemic Clamp Trial to Evaluate Pharmacokinetics of Single Doses of BioChaperone Insulin Lispro in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BC3-CT017
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- BioChaperone insulin lispro 0.1 U/kg (Experimental)
  Interventions: Drug: Biochaperone insulin lispro 0.1 U/kg
- BioChaperone insulin lispro 0.2 U/kg (Experimental)
  Interventions: Drug: Biochaperone insulin lispro 0.2 U/kg
- BioChaperone insulin lispro 0.4 U/kg (Experimental)
  Interventions: Drug: Biochaperone insulin lispro 0.4 U/kg
- Humalog® (Active Comparator)
  Interventions: Drug: Humalog®

INTERVENTIONS:
Drug: Biochaperone insulin lispro 0.1 U/kg — Injection of a single dose of BioChaperone insulin lispro at the dose of 0.1 U/kg
  Arms: BioChaperone insulin lispro 0.1 U/kg
Drug: Biochaperone insulin lispro 0.2 U/kg — Injection of a single dose of BioChaperone insulin lispro at the dose of 0.2 U/kg
  Arms: BioChaperone insulin lispro 0.2 U/kg
Drug: Biochaperone insulin lispro 0.4 U/kg — Injection of a single dose of BioChaperone insulin lispro at the dose of 0.4 U/kg
  Arms: BioChaperone insulin lispro 0.4 U/kg
Drug: Humalog® — Injection of a single dose of Humalog® at the dose of 0.2 U/kg
  Arms: Humalog®

SUMMARY:
This is a double-blind, randomised, three period crossover phase 1 trial using automated 8-hour euglycemic clamps in healthy Japanese subjects.

Each subject will be randomly allocated to one out of nine sequences to receive either three single doses of BioChaperone insulin lispro or one single dose of Humalog® and two single doses of BioChaperone insulin lispro on three separate dosing visits.

The total trial maximum duration for a subject will be up to 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male or female subjects by completion of medical history, physical examination and biochemical investigations as judged by the Investigator.
* BMI between 18.5 and 25.0 kg∙m-2, both inclusive.
* Fasting Plasma Glucose ≤ 5.6 mmol/L (100 mg/dL).
* Signed and dated informed consent obtained before any trial-related activities.

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products.
* Receipt of any investigational medicinal product within 3 months before randomisation in this trial.
* Any history or presence of a life threatening disease (i.e. cancer except basal cell skin cancer or squamous cell skin cancer), or of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic (including type 1 and type 2 diabetes mellitus, haematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynaecologic (if female), or infectious disease, or signs of acute illness as judged by the investigator.
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
AUCLispro(0-30min) | Up to 30 minutes
  Area under the insulin lispro serum concentration - time curve from t=0 to 30 minutes

SECONDARY OUTCOMES:
AUCGIR(0-last) | Up to 8 hours
  Area under the glucose infusion rate time curve from 0 hours until the end of clamp
Adverse Events | Up to 10 weeks
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — Profil GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany